CLINICAL TRIAL: NCT01597245
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Comparing the Efficacy and Safety of LY2439821 to Etanercept and Placebo in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Phase 3 Study in Participants With Moderate to Severe Psoriasis (UNCOVER-2)
Acronym: UNCOVER-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12973; I1F-MC-RHBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2020-06-26 (Actual); Status verified 2019-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — ixekizumab; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 80 mg ixekizumab Dosing Regimen 1 (Experimental): Administered by two 80 mg subcutaneous (SC) injections at Week 0, then one 80 mg SC injection per Dosing Regimen 1 until Week 12. At Week 12, ixekizumab responders are re-randomized to placebo, Dosing Regimen 2 or Dosing Regimen 3. Ixekizumab non-responders are assigned to Dosing Regimen 2.
  Interventions: Drug: 80 mg ixekizumab Dosing Regimen
- 80 mg ixekizumab Dosing Regimen 2 (Experimental): Administered by two 80 mg SC injections at Week 0, then one 80 mg SC injection per Dosing Regimen 2 until Week 12. At Week 12, ixekizumab responders are re-randomized to placebo, Dosing Regimen 2 or Dosing Regimen 3. Ixekizumab non-responders are assigned to Dosing Regimen 2.
  Interventions: Drug: 80 mg ixekizumab Dosing Regimen
- 80 mg ixekizumab Dosing Regimen 3 (Experimental): Dosing Regimen 3 is not used until Week 12. At Week 12, ixekizumab responders re-randomized to this arm will receive Dosing Regimen 3.
  Interventions: Drug: 80 mg ixekizumab Dosing Regimen
- 50 mg etanercept (Active Comparator): Administered by one 50 mg SC injection twice weekly starting at Week 0 up to Week 12. At Week 12, etanercept responders are assigned to placebo, and nonresponders to Dosing Regimen 2.
  Interventions: Drug: 50 mg etanercept
- Placebo for ixekizumab (Placebo Comparator): Placebo for ixekizumab administered by two SC injections at Week 0, then one SC injection per Dosing Regimen 1 until Week 12. At Week 12, placebo responders are assigned to placebo, and nonresponders to Dosing Regimen 2. Placebo for etanercept administered by one SC injection twice weekly starting at Week 0 up to Week 12 was used to blind etanercept injections for Dosing Regimen 1, Dosing Regimen 2, and Placebo Comparator groups.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 80 mg ixekizumab Dosing Regimen — Administered SC
  Other Names: LY2439821
  Arms: 80 mg ixekizumab Dosing Regimen 1; 80 mg ixekizumab Dosing Regimen 2; 80 mg ixekizumab Dosing Regimen 3
Drug: 50 mg etanercept — Administered SC
  Arms: 50 mg etanercept
Drug: Placebo — Administered SC
  Arms: Placebo for ixekizumab

SUMMARY:
This study will assess the safety and efficacy of ixekizumab (LY2439821) compared to etanercept and placebo in participants with moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Present with chronic plaque psoriasis based on a confirmed diagnosis of chronic plaque psoriasis for at least 6 months prior to first dose of study drug
* At least 10% Body Surface Area (BSA) of psoriasis at screening and at first dose of study drug
* Static Physician Global Assessment (sPGA) score of at least 3 and Psoriasis Area and Severity Index (PASI) score of at least 12 at screening and at first dose of study drug
* Candidate for phototherapy and/or systemic therapy
* Men must agree to use a reliable method of birth control or remain abstinent during the study
* Women must agree to use reliable birth control or remain abstinent during the study and for at least 12 weeks after stopping treatment

Exclusion Criteria:

* Pustular, erythrodermic, and/or guttate forms of psoriasis
* History of drug-induced psoriasis
* Prior use of etanercept
* Clinically significant flare of psoriasis during the 12 weeks prior to randomization
* Concurrent or recent use of any biologic agent
* Received non-biologic systemic psoriasis therapy or phototherapy (including psoralens and ultraviolet A [PUVA], ultraviolet B [UVB]) within the previous 4 weeks; or had topical psoriasis treatment within the previous 2 weeks prior to randomization
* Cannot avoid excessive sun exposure or use of tanning booths for at least 4 weeks prior to randomization and during the study
* Have participated in any study with interleukin 17 (IL-17) antagonists, including ixekizumab
* Serious disorder or illness other than plaque psoriasis
* Serious infection within the last 3 months
* Breastfeeding or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1224 (Actual)
Dates: Start 2012-05-18 (Actual); Primary Completion 2014-03-25 (Actual); Study Completion 2019-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (118):
- United States (41):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Riverside, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Farmington, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boca Raton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeLand, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., West Palm Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alpharetta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plainfield, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Overland Park, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baton Rouge, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Silver Spring, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Andover, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Worcester, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paramus, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Verona, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wilmington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norman, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greer, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bristol, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Webster, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norfolk, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington
- Australia (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phillip, Australian Capital Territory
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Leonards, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sydney, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Woolloogabba, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hectorville, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Box Hill, Victoria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carlton, Victoria
- Austria (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Feldkirch
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Innsbruck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Canada (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Surrey, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barrie, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamilton, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Markham, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Bay, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peterborough, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sainte-Foy, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
- Czechia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Prague
- France (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Amiens
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Besançon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boulogne
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cannes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chambray-lès-Tours
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nice
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paris
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poitiers
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rouen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Darmstadt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dresden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Essen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Giessen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Göttingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osnabrück
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tübingen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Witten
- Netherlands (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Breda
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nijmegen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam
- Poland (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gdansk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kielce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lodz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Opole
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Craiova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iași
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timișoara
- Spain (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alcorcón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alicante
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Badalona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Palmas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- United Kingdom (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dundee, Angus
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Hampstead
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glasgow, Scotland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lanarkshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salford
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scunthorpe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Plan Description:
  Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org

REFERENCES:
- [Derived] Egeberg A, Hawkes JE, Somani N, Burge R, See K, Gallo G, McKean-Matthews M, Gooderham M, Han G, Armstrong A. Sustained Improvements in Clinical and Patient-Reported Outcomes and Quality of Life Through 5 Years Among Ixekizumab-Treated Patients with Complete Clearance of Scalp Psoriasis by Week 60. Dermatol Ther (Heidelb). 2024 Apr;14(4):1007-1018. doi: 10.1007/s13555-024-01147-7. Epub 2024 Apr 22. PMID 38647975
- [Derived] Armstrong A, Gonzalez-Cantero A, Khattri S, Muzy G, Malatestinic WN, Lampropoulou A, Feely M, See SK, Mert C, Blauvelt A. Comparing Achievement of National Psoriasis Foundation Treatment Targets among Patients with Plaque Psoriasis Treated with Ixekizumab versus Other Biologics in Clinical and Real-World Studies. Dermatol Ther (Heidelb). 2024 Apr;14(4):933-952. doi: 10.1007/s13555-024-01136-w. Epub 2024 Mar 23. PMID 38521874
- [Derived] Kirkham BW, Egeberg A, Behrens F, Pinter A, Merola JF, Holzkamper T, Gallo G, Ng KJ, Bolce R, Schuster C, Nash P, Puig L. A Comprehensive Review of Ixekizumab Efficacy in Nail Psoriasis from Clinical Trials for Moderate-to-Severe Psoriasis and Psoriatic Arthritis. Rheumatol Ther. 2023 Oct;10(5):1127-1146. doi: 10.1007/s40744-023-00553-1. Epub 2023 Jul 3. PMID 37400681
- [Derived] Elewski BE, Blauvelt A, Gallo G, Wolf E, McKean-Matthews M, Burge R, Merola JF, Gottlieb AB, Guenther LC. Simultaneous Nail and Skin Clearance in Ixekizumab Head-to-Head Trials for Moderate-to-Severe Psoriasis and Psoriatic Arthritis. Dermatol Ther (Heidelb). 2022 Apr;12(4):911-920. doi: 10.1007/s13555-022-00704-2. Epub 2022 Mar 13. PMID 35279805
- [Derived] Rich P, Goldblum O, Disch D, Lin CY, Merola JF, Elewski B. Nail Psoriasis Does Not Affect Skin Response to Ixekizumab in Patients With Moderate-To-Severe Psoriasis. J Drugs Dermatol. 2020 Aug 1;19(8):741-746. doi: 10.36849/JDD.2020.5116. PMID 32845588
- [Derived] Leonardi C, Reich K, Foley P, Torii H, Gerdes S, Guenther L, Gooderham M, Ferris LK, Griffiths CEM, ElMaraghy H, Crane H, Patel H, Burge R, Gallo G, Shrom D, Leung A, Lin CY, Papp K. Efficacy and Safety of Ixekizumab Through 5 Years in Moderate-to-Severe Psoriasis: Long-Term Results from the UNCOVER-1 and UNCOVER-2 Phase-3 Randomized Controlled Trials. Dermatol Ther (Heidelb). 2020 Jun;10(3):431-447. doi: 10.1007/s13555-020-00367-x. Epub 2020 Mar 21. PMID 32200512
- [Derived] Yosipovitch G, Reich A, Steinhoff M, Beselin A, Kent T, Dossenbach M, Berggren L, Henneges C, Luger T. Impact of Ixekizumab Treatment on Itch and Psoriasis Area and Severity Index in Patients with Moderate-to-Severe Plaque Psoriasis: An Integrated Analysis of Two Phase III Randomized Studies. Dermatol Ther (Heidelb). 2018 Dec;8(4):621-637. doi: 10.1007/s13555-018-0267-9. Epub 2018 Nov 21. PMID 30465321
- [Derived] Blauvelt A, Papp KA, Griffiths CEM, Puig L, Weisman J, Dutronc Y, Kerr LF, Ilo D, Mallbris L, Augustin M. Efficacy and Safety of Switching to Ixekizumab in Etanercept Non-Responders: A Subanalysis from Two Phase III Randomized Clinical Trials in Moderate-to-Severe Plaque Psoriasis (UNCOVER-2 and -3). Am J Clin Dermatol. 2017 Apr;18(2):273-280. doi: 10.1007/s40257-016-0246-9. PMID 28074446
- [Derived] Gordon KB, Blauvelt A, Papp KA, Langley RG, Luger T, Ohtsuki M, Reich K, Amato D, Ball SG, Braun DK, Cameron GS, Erickson J, Konrad RJ, Muram TM, Nickoloff BJ, Osuntokun OO, Secrest RJ, Zhao F, Mallbris L, Leonardi CL; UNCOVER-1 Study Group; UNCOVER-2 Study Group; UNCOVER-3 Study Group. Phase 3 Trials of Ixekizumab in Moderate-to-Severe Plaque Psoriasis. N Engl J Med. 2016 Jul 28;375(4):345-56. doi: 10.1056/NEJMoa1512711. Epub 2016 Jun 8. PMID 27299809
- [Derived] Armstrong AW, Lynde CW, McBride SR, Stahle M, Edson-Heredia E, Zhu B, Amato D, Nikai E, Yang FE, Gordon KB. Effect of Ixekizumab Treatment on Work Productivity for Patients With Moderate-to-Severe Plaque Psoriasis: Analysis of Results From 3 Randomized Phase 3 Clinical Trials. JAMA Dermatol. 2016 Jun 1;152(6):661-9. doi: 10.1001/jamadermatol.2016.0269. PMID 26953848
- [Derived] Griffiths CE, Reich K, Lebwohl M, van de Kerkhof P, Paul C, Menter A, Cameron GS, Erickson J, Zhang L, Secrest RJ, Ball S, Braun DK, Osuntokun OO, Heffernan MP, Nickoloff BJ, Papp K; UNCOVER-2 and UNCOVER-3 investigators. Comparison of ixekizumab with etanercept or placebo in moderate-to-severe psoriasis (UNCOVER-2 and UNCOVER-3): results from two phase 3 randomised trials. Lancet. 2015 Aug 8;386(9993):541-51. doi: 10.1016/S0140-6736(15)60125-8. Epub 2015 Jun 10. PMID 26072109

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study has 5 periods: Period 1 - Screening; Period 2 - Blinded Induction Dosing Period (Weeks 0 to 12); Period 3 - Blinded Maintenance Dosing Period (Weeks 12 - 60); Period 4 - Long-Term Extension Period (Weeks 60 - 264); Period 5 - Post-Treatment Follow-Up Period (A Minimum of 12 Weeks)
Groups:
- Placebo- Induction Period: Placebo was administered as 2 subcutaneous (SC) injections at week 0, followed by 1 injection at weeks 2, 4, 6, 8, 10. Placebo for ETN (1 SC injection) administered twice weekly (every 3 to 4 days) starting at Week 0 up to Week 12.
- 50 mg Etanercept (ETN) - Induction Period: 50 milligrams (mg) ETN was administered by 1 SC injection twice weekly (every 3-4 days) up to Week 12. Placebo for ixe was administered as 2 SC injections at Week 0 followed by Placebo for ixe administered as 1 SC injection Q2W (Weeks 2, 4, 6, 8, and 10).
- Ixe Q4W - Induction Period: 160 mg ixekizumab (ixe) was administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection every 4 weeks (Q4W:Weeks 4 and 8). Placebo was administered as 1 SC injection at Weeks 2, 6, and 10. Placebo for ETN (1 SC injection) was administered twice weekly starting at Week 0 up to Week 12.
- Ixe Q2W - Induction Period: 160 mg ixe administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection Q2W at Weeks 2, 4, 6, 8, and 10. Placebo for ETN (1 SC injection) was administered twice weekly starting at Week 0 up to Week 12
- Ixe/Placebo- Maintenance Period Primary Population (Pop): Participants who received 80 mg ixe Q2W or Q4W in Induction Period (Weeks 0 to 10) and classified as responders were administered placebo as 2 SC injections at Week 12 followed by placebo as 1 SC injection Q4W up to and including Week 56.
- Ixe/Ixe Q4W - Maintenance Period Primary Pop: Participants who received 80 mg ixe Q2W or Q4W in Induction Period (Weeks 0 to 10) and classified as responders were administered 80 mg ixe as 1 SC injection and a Placebo for ixe injection at Week 12 followed by 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- Ixe/Ixe Q12W - Maintenance Period Primary Pop: Participants who received 80 mg ixe Q2W or Q4W in Induction Period (Weeks 0 to 10) and classified as responders were administered 80 mg ixe as 1 SC injection and a Placebo for ixe injection at Week 12 followed by 80 mg ixe as 1 SC injection every 12 weeks (Q12W) up to and including Week 56. To maintain blinding with Q4W dose regimen, Placebo for ixe given as 1 SC injection at Weeks 16, 20, 28, 32, 40, 44, 52, and 56.
- Placebo Resp/Placebo - Maintenance Period Secondary Pop: Participants who received placebo during the Induction Period (Weeks 0 to 10) and classified as responders (resp) and were administered placebo as 2 SC injections at Week 12 followed by placebo as 1 SC injection Q4W up to and including Week 56.
- Placebo NonResp/Ixe Q4W - Maintenance Period Secondary Pop: Participants who received placebo in Induction Period (Weeks 0 to 10) and classified as non-responders (NonResp) were administered 160 mg ixe as 2 SC injections at Week 12 followed by 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- ETN Resp/Placebo Maintenance Period Secondary Pop: Participants who received ETN during the Induction Period (Weeks 0 to 10) and classified as responders and were administered placebo as 2 SC injections at Week 12 followed by placebo as 1 SC injection Q4W up to and including Week 56.
- ETN NonResp/Ixe Q4W - Maintenance Period Secondary Pop: Participants who received ETN in Induction Period (Weeks 0 to 12) and classified as non-responders were administered 2 SC injections of placebo at Week 12 followed by 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- Ixe Q4W NonResp/Ixe Q4W - Maintenance Period Secondary Pop: Participants who received 80 mg ixe Q4W in Induction Period (Weeks 0 to 10) and classified as non-responders were administered 80 mg ixe as 1 SC injection and a Placebo for ixe injection at Week 12 followed by 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- Ixe Q2W NonResp/Ixe Q4W - Maintenance Period Secondary Pop: Participants who received 80 mg ixe Q2W in Induction Period (Weeks 0 to 10) and classified as non-responders were administered 80 mg ixe as 1 SC injection and a Placebo for ixe injection at Week 12 followed by 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- Placebo Long-Term Extension (LTE): Participants who received placebo at the start of long-term extension period (Week 60) and could be switched to ixe. Data while participants were on placebo were included.
- Ixe Long-Term Extension: Participants who received 80 mg ixe in all dosing regimens at the start of the long-term extension period from Week 60 to Week 264.
- Total Ixe Long-Term Extension: Participants who received at least 1 dose of 80 mg ixe in all dosing regimens during the long-term extension period from Week 60 to Week 264, including those who have switched from PBO to Ixe in long-term extension (LTE) period.
- Placebo Post-Treatment Follow-Up: Participants who received PBO immediately prior to entering the Post-Treatment Follow-Up period (a 12-24 week period after their last scheduled treatment visit).
- ETN Post-Treatment Follow-Up: Participants who received ETN immediately prior to entering the Post-Treatment Follow-Up period (a 12-24 week period after their last scheduled treatment visit).
- Ixe Q12W Post-Treatment Follow-Up: Participants who received 80 mg ixe 1 SC injection Q12W immediately prior to entering the Post-Treatment Follow-Up period (a 12-24 week period after their last scheduled treatment visit).
- Ixe Q4W Post-Treatment Follow-Up: Participants who received 80 mg ixe 1 SC injection Q4W immediately prior to entering the Post-Treatment Follow-Up period (a 12-24 week period after their last scheduled treatment visit).
- Ixe Q2W Post-Treatment Follow-Up: Participants who received 80 mg ixe 1 SC injection Q2W immediately prior to entering the Post-Treatment Follow-Up period (a 12-24 week period after their last scheduled treatment visit).
Period: Induction Period (Week 0 - Week 12)
Arm/Group | Placebo- Induction Period | 50 mg Etanercept (ETN) - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period | Ixe/Placebo- Maintenance Period Primary Population (Pop) | Ixe/Ixe Q4W - Maintenance Period Primary Pop | Ixe/Ixe Q12W - Maintenance Period Primary Pop | Placebo Resp/Placebo - Maintenance Period Secondary Pop | Placebo NonResp/Ixe Q4W - Maintenance Period Secondary Pop | ETN Resp/Placebo Maintenance Period Secondary Pop | ETN NonResp/Ixe Q4W - Maintenance Period Secondary Pop | Ixe Q4W NonResp/Ixe Q4W - Maintenance Period Secondary Pop | Ixe Q2W NonResp/Ixe Q4W - Maintenance Period Secondary Pop | Placebo Long-Term Extension (LTE) | Ixe Long-Term Extension | Total Ixe Long-Term Extension | Placebo Post-Treatment Follow-Up | ETN Post-Treatment Follow-Up | Ixe Q12W Post-Treatment Follow-Up | Ixe Q4W Post-Treatment Follow-Up | Ixe Q2W Post-Treatment Follow-Up
Started | 168 | 358 | 347 | 351 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 167 | 357 | 347 | 350 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 158 | 333 (1 participant randomized to maintenance period but did not receive a dose in the maintenance period.) | 328 | 342 (2 participants discontinued after IND completion and prior to randomizing into maintenance period.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 25 | 19 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 5 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 8 | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 4 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Period (Week 12 to Week 60)
Arm/Group | Placebo- Induction Period | 50 mg Etanercept (ETN) - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period | Ixe/Placebo- Maintenance Period Primary Population (Pop) | Ixe/Ixe Q4W - Maintenance Period Primary Pop | Ixe/Ixe Q12W - Maintenance Period Primary Pop | Placebo Resp/Placebo - Maintenance Period Secondary Pop | Placebo NonResp/Ixe Q4W - Maintenance Period Secondary Pop | ETN Resp/Placebo Maintenance Period Secondary Pop | ETN NonResp/Ixe Q4W - Maintenance Period Secondary Pop | Ixe Q4W NonResp/Ixe Q4W - Maintenance Period Secondary Pop | Ixe Q2W NonResp/Ixe Q4W - Maintenance Period Secondary Pop | Placebo Long-Term Extension (LTE) | Ixe Long-Term Extension | Total Ixe Long-Term Extension | Placebo Post-Treatment Follow-Up | ETN Post-Treatment Follow-Up | Ixe Q12W Post-Treatment Follow-Up | Ixe Q4W Post-Treatment Follow-Up | Ixe Q2W Post-Treatment Follow-Up
Started | 0 (Participants who completed the prior period and then randomized to the maintenance period.) | 0 (Participants who completed the prior period and then randomized to the maintenance period.) | 0 (Participants who completed the prior period and then randomized to the maintenance period.) | 0 (Participants who completed the prior period and then randomized to the maintenance period.) | 176 (Participants who completed the prior period and then randomized to the maintenance period.) | 187 (Participants who completed the prior period and then randomized to the maintenance period.) | 181 (Participants who completed the prior period and then randomized to the maintenance period.) | 3 (Participants who completed the prior period and then randomized to the maintenance period.) | 155 (Participants who completed the prior period and then randomized to the maintenance period.) | 132 (Participants who completed the prior period and then randomized to the maintenance period.) | 200 (Participants who completed the prior period and then randomized to the maintenance period.) | 75 (Participants who completed the prior period and then randomized to the maintenance period.) | 49 (Participants who completed the prior period and then randomized to the maintenance period.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Participants Received One Dose | 0 | 0 | 0 | 0 | 176 | 187 | 181 | 3 | 155 | 132 | 200 | 75 | 49 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 15 | 149 | 92 | 0 | 135 | 11 | 178 | 56 | 37 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 161 | 38 | 89 | 3 | 20 | 121 | 22 | 19 | 12 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — On study treatment | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Relapsed | 0 | 0 | 0 | 0 | 150 | 22 | 80 | 2 | 0 | 114 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 2 | 10 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 4 | 6 | 6 | 1 | 8 | 2 | 8 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 0 | 4 | 1 | 6 | 5 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 3 | 4 | 1 | 0 | 1 | 2 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Long Term Extension (Week 60 - Week 264)
Arm/Group | Placebo- Induction Period | 50 mg Etanercept (ETN) - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period | Ixe/Placebo- Maintenance Period Primary Population (Pop) | Ixe/Ixe Q4W - Maintenance Period Primary Pop | Ixe/Ixe Q12W - Maintenance Period Primary Pop | Placebo Resp/Placebo - Maintenance Period Secondary Pop | Placebo NonResp/Ixe Q4W - Maintenance Period Secondary Pop | ETN Resp/Placebo Maintenance Period Secondary Pop | ETN NonResp/Ixe Q4W - Maintenance Period Secondary Pop | Ixe Q4W NonResp/Ixe Q4W - Maintenance Period Secondary Pop | Ixe Q2W NonResp/Ixe Q4W - Maintenance Period Secondary Pop | Placebo Long-Term Extension (LTE) | Ixe Long-Term Extension | Total Ixe Long-Term Extension | Placebo Post-Treatment Follow-Up | ETN Post-Treatment Follow-Up | Ixe Q12W Post-Treatment Follow-Up | Ixe Q4W Post-Treatment Follow-Up | Ixe Q2W Post-Treatment Follow-Up
Started | 0 | 0 | 0 | 0 | 0 (Includes participants who started the long-term extension period.) | 0 (Includes participants who started the long-term extension period.) | 0 (Includes participants who started the long-term extension period.) | 0 | 0 (Includes participants who started the long-term extension period.) | 0 (Includes participants who started the long-term extension period.) | 0 (Includes participants who started the long-term extension period.) | 0 (Includes participants who started the long-term extension period.) | 0 (Includes participants who started the long-term extension period.) | 26 (Participants who received placebo at the start of the long-term extension period.) | 979 (Participants received ixe at the start of the long-term extension.) | 1002 (Participants received ixe in all dosing regimens, including participants who switched PBO to ixe.) | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 754 | 774 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 225 | 228 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 69 | 70 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 62 | 63 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 38 | 38 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 26 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 11 | 12 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical Relapse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Switched from PBO to Ixe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Post Treatment Follow-Up (12 - 24 Weeks)
Arm/Group | Placebo- Induction Period | 50 mg Etanercept (ETN) - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period | Ixe/Placebo- Maintenance Period Primary Population (Pop) | Ixe/Ixe Q4W - Maintenance Period Primary Pop | Ixe/Ixe Q12W - Maintenance Period Primary Pop | Placebo Resp/Placebo - Maintenance Period Secondary Pop | Placebo NonResp/Ixe Q4W - Maintenance Period Secondary Pop | ETN Resp/Placebo Maintenance Period Secondary Pop | ETN NonResp/Ixe Q4W - Maintenance Period Secondary Pop | Ixe Q4W NonResp/Ixe Q4W - Maintenance Period Secondary Pop | Ixe Q2W NonResp/Ixe Q4W - Maintenance Period Secondary Pop | Placebo Long-Term Extension (LTE) | Ixe Long-Term Extension | Total Ixe Long-Term Extension | Placebo Post-Treatment Follow-Up | ETN Post-Treatment Follow-Up | Ixe Q12W Post-Treatment Follow-Up | Ixe Q4W Post-Treatment Follow-Up | Ixe Q2W Post-Treatment Follow-Up
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (Participants who completed or discontinued from study treatment and entered the follow-up period.) | 0 (Participants who completed or discontinued from study treatment and entered the follow-up period.) | 16 (Participants who completed or discontinued from study treatment and entered the follow-up period.) | 6 (Participants who completed or discontinued from study treatment and entered the follow-up period.) | 24 (Participants who completed or discontinued from study treatment and entered the follow-up period.) | 656 (Participants who completed or discontinued from study treatment and entered the follow-up period.) | 248 (Participants who completed or discontinued from study treatment and entered the follow-up period.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 489 | 212
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 6 | 10 | 167 | 36
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 5 | 8 | 63 | 13
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 41 | 13
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 29 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 14 | 4
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 9 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 6 | 2
Not completed — Entry Criteria Not Met | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Clinical Relapse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo - Induction Period: Placebo was administered as 2 subcutaneous (SC) injections at week 0, followed by 1 injection at weeks 2, 4, 6, 8, 10. Placebo for ETN (1 SC injection) administered twice weekly (every 3 to 4 days) starting at Week 0 up to Week 12.
- 50 mg ETN - Induction Period: 50 mg ETN was administered by 1 SC injection twice weekly (every 3-4 days) up to Week 12. Placebo for ixe was administered as 2 SC injections at Week 0 followed by Placebo for ixe administered as 1 SC injection Q2W (Weeks 2, 4, 6, 8, and 10).
- Ixe Q4W - Induction Period: 160 mg ixe was administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection every 4 weeks (Q4W: Weeks 4 and 8). Placebo was administered as 1 SC injection at Weeks 2, 6, and 10. Placebo for ETN (1 SC injection) was administered twice weekly starting at Week 0 up to Week 12.
- Total: Total of all reporting groups
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period | Total
Number analyzed (Participants) | 168 | 358 | 347 | 351 | 1224
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 159 | 337 | 324 | 327 | 1147
  >=65 years | 9 | 21 | 23 | 24 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 122 | 103 | 130 | 403
  Male | 120 | 236 | 244 | 221 | 821
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 26 | 24 | 19 | 80
  Not Hispanic or Latino | 130 | 279 | 271 | 274 | 954
  Unknown or Not Reported | 27 | 53 | 52 | 58 | 190
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2 | 2 | 6
  Asian | 6 | 8 | 11 | 12 | 37
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 0 | 3
  Black or African American | 10 | 13 | 11 | 5 | 39
  White | 149 | 331 | 315 | 330 | 1125
  More than one race | 0 | 1 | 3 | 1 | 5
  Unknown or Not Reported | 0 | 4 | 4 | 1 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 40 | 82 | 82 | 84 | 288
  Austria | 2 | 10 | 6 | 5 | 23
  Netherlands | 1 | 2 | 2 | 1 | 6
  Czechia | 3 | 6 | 3 | 6 | 18
  Romania | 6 | 9 | 8 | 12 | 35
  United States | 49 | 111 | 105 | 104 | 369
  Poland | 14 | 30 | 28 | 30 | 102
  United Kingdom | 4 | 9 | 9 | 11 | 33
  Australia | 7 | 13 | 15 | 16 | 51
  France | 7 | 18 | 21 | 19 | 65
  Germany | 28 | 53 | 51 | 47 | 179
  Spain | 7 | 15 | 17 | 16 | 55
Baseline in Static Physician Global Assessment (sPGA) [Count of Participants; unit: Participants] — The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. The sPGA is recommended as an endpoint to use to assess efficacy in the treatment of Ps (EMEA 2004). Overall lesions are categorized by descriptions for induration, erythema, and scaling. For the analysis of responses, the participant's Ps is assessed at a given time point on a 6-point scale in which 0 = cleared, 1 = minimal, 2 = mild, 3 = moderate; 4 = severe, 5 = very severe.
  Participants
    sPGA = 3 | 86 | 186 | 166 | 178 | 616
    sPGA = 4,5 | 82 | 172 | 181 | 173 | 608
Baseline in Participants Achieving Psoriasis Area and Severity Index (PASI) Score [Mean (Standard Deviation); unit: units on a scale] — PASI is another accepted primary efficacy measurement for this phase of development of Ps treatments. The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation, erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 or no Ps to 72 for the most severe disease.
  units on a scale | 20.57 (8.366) | 19.07 (6.701) | 20.04 (6.962) | 19.35 (7.339) | 19.63 (7.216)
Baseline Dermatology-Specific Quality of Life Index (DLQI) Total Score [Mean (Standard Deviation); unit: units on a scale] — DLQI is a participant-administered, 10-question, validated, quality-of-life questionnaire that covers 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include 0 (not at all), 1 (a little), 2 (a lot), and 3 (very much) and unanswered ("not relevant") responses were scored as "0." Total scores range from 0 to 30, with higher score indicating greater quality of life impairment.
  units on a scale | 12.8 (7.24) | 12.7 (7.03) | 11.6 (6.65) | 12.4 (6.86) | 12.3 (6.91)
Baseline in Nail Psoriasis Severity Index (NAPSI) Total Score [Mean (Standard Deviation); unit: units on a scale] — The NAPSI scale evaluates Ps severity in the fingernail bed and fingernail matrix with each divided into quadrants. Scores range from 0 (none) to 4 (Ps in all 4 quadrants), depending on the presence (score of 1) or absence (score of 0) of Ps in each quadrant of the fingernail bed or matrix. NAPSI score of a fingernail is the sum of scores from each quadrant of the fingernail bed and fingernail matrix (maximum of 8). The total NAPSI score equals the sum of all fingernails and ranges from 0 to 80. Higher scores indicate more severe Ps.
  units on a scale | 27.62 (20.937) | 30.44 (20.648) | 23.70 (18.696) | 26.27 (20.388) | 26.97 (20.211)
Baseline in Psoriasis Scalp Severity Index (PSSI) Total Score [Mean (Standard Deviation); unit: units on a scale] — The PSSI is a physician assessment of erythema, induration and desquamation and percent of scalp that is covered with a scores range from 0 (none) to 4 (very severe). The composite score is derived from the sum of scores for erythema, induration, and desquamation multiplied by the score recorded for the extent of the scalp area involved, 1 (<10%) to 6 (90%-100%) with a total score ranging from 0 (less severity) to 72 (more severity).
  units on a scale | 21.0 (15.24) | 20.0 (15.19) | 20.8 (15.63) | 19.5 (14.85) | 20.2 (15.22)
Baseline in Body Surface Area (BSA) Total Score [Mean (Standard Deviation); unit: units on a scale] — BSA is a physician rating of the percentage of involvement of Ps for each participant. BSA is assessed on a continuous scale from 0% (no involvement) to 100% (full involvement), where 1% corresponds to the size of the participant's hand (includes the palm, fingers and thumb). Total BSA is the sum of handprints from the affected areas.
  units on a scale | 27.2 (18.12) | 25.3 (15.50) | 27.0 (17.23) | 25.1 (15.82) | 26.0 (16.47)
Baseline in Quick Inventory of Depressive Symptomatology Self Report 16 items (QIDS-SR16) Score [Mean (Standard Deviation); unit: units on a scale] — QIDS-SR16 is a participant-administered, 16-item instrument assesses the existence and severity of symptoms of depression. A participant is asked a statement relating to the way they have felt for the past 7 days and rate on a 4-point scale: 0 (best) to 3 (worst). The sum of the domains [sad mood, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, sleep disturbance, decrease/increase in appetite/weight, and psychomotor agitation/retardation] to give a single total scores range from 0 to 27, with higher scores indicating greater symptom severity.
  units on a scale | 4.7 (4.14) | 4.5 (4.07) | 4.4 (4.04) | 4.6 (3.84) | 4.5 (4.00)
Baseline in Work Productivity Activity Impairment Questionnaire-Psoriasis (WPAI-PSO) Total Score [Mean (Standard Deviation); unit: units on a scale] — The (WPAI-PSO) is a 6-item instrument to assess the impact of psoriasis on productivity impairment within the past 7 days and has four domains: absenteeism, presenteeism (reduced productivity while at work), an overall work impairment score, and impairment in daily activities performed outside of work. Four scores are derived as percentages: absenteeism, presenteeism, overall work impairment (absenteeism and presenteeism), and impairment in activities performed outside of work. Percentage is calculated as each score * 100 and ranges from 0-100; greater scores indicate greater impairment.
  units on a scale
    Absenteeism Score | 4.3 (16.61) | 3.7 (15.24) | 4.6 (17.65) | 7.3 (22.15) | 5.1 (18.40)
    Active Impairment Score | 30.2 (28.87) | 31.3 (29.04) | 29.4 (29.28) | 31.7 (29.64) | 30.7 (29.24)
    Presenteeism Score | 24.3 (26.19) | 21.2 (25.42) | 22.3 (24.77) | 24.2 (25.80) | 22.8 (25.44)
    Work Productivity Loss | 26.1 (28.11) | 22.3 (26.52) | 24.6 (27.41) | 27.7 (29.19) | 25.0 (27.82)
Baseline in Short form (36 Items) Health Survey SF-36 Total Score [Mean (Standard Deviation); unit: units on a scale] — The SF-36 is a self-reported instrument that measures the participant's health status during the previous 7 days. It comprises 36-items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. The 8 domains are regrouped in the Physical Component Score (PCS) and Mental Component Score (MCS) scores. Scores range from 0 to 100, with higher scores indicating better levels of function and/or better health.
  units on a scale
    Physical Summary Score | 47.7094 (9.5043) | 47.5268 (9.0729) | 47.6231 (8.9693) | 47.6996 (9.0332) | 47.6289 (9.0814)
    Mental Summary Score | 47.7889 (10.6183) | 48.7097 (10.6546) | 49.0131 (10.9087) | 47.7140 (11.6686) | 48.3832 (11.0234)
Baseline in Patient's Global Assessment (PatGA) Total Score [Mean (Standard Deviation); unit: units on a scale] — The PatGA is a single-item self-reported instrument asking the participant to rate the severity of their psoriasis "today" by circling a number on the numeric rating scale from 0 (Clear = no psoriasis) to 5 (Severe = the worst their psoriasis has ever been).
  units on a scale | 4.0 (0.92) | 4.0 (0.96) | 4.1 (0.90) | 4.1 (0.91) | 4.0 (0.92)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Static Physician Global Assessment (sPGA) of (0,1) (Efficacy of Ixekizumab in Participants With Moderate to Severe Chronic Plaque Psoriasis. Measure: Static Physician Global Assessment [sPGA])
Description: The sPGA is the physician's determination of the participant's Psoriasis (Ps) lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participant's Ps was assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe). An sPGA responder was defined as having a post-baseline sPGA score of "0" or "1" with at least a 2-point improvement from baseline.
Time Frame: Week 12
Population: All randomized participants. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: percentage of participants
Groups:
- 50 mg Etanercept (ETN) - Induction Period: 50 mg ETN was administered by 1 SC injection twice weekly (every 3-4 days) up to Week 12. Placebo for ixe was administered as 2 SC injections at Week 0 followed by Placebo for ixe administered as 1 SC injection Q2W (Weeks 2, 4, 6, 8, and 10).
Arm/Group | Placebo - Induction Period | 50 mg Etanercept (ETN) - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 168 | 358 | 347 | 351
percentage of participants | 2.4 | 36.0 | 72.9 | 83.2
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg Etanercept (ETN) - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

2. Primary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) ≥75% (PASI75) Improvement (Efficacy of Ixekizumab in Participants With Moderate to Severe Chronic Plaque Psoriasis. Measure: Psoriasis Area and Severity Index [PASI])
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored separately and the scores then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor (head [0.1], upper limbs [0.2], trunk [0.3], lower limbs [0.4]). Overall scores range from 0 (no Ps) to 72 (the most severe disease). Participants achieving PASI75 were defined as having an improvement of ≥75% in the PASI score compared to baseline.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Ixe Q4W - Induction Period: 160 mg ixe was administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection every 4 weeks (Q4W; Weeks 4 and 8). Placebo was administered as 1 SC injection at Weeks 2, 6, and 10. Placebo for ETN (1 SC injection) was administered twice weekly starting at Week 0 up to Week 12.
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 168 | 358 | 347 | 351
percentage of participants | 2.4 | 41.6 | 77.5 | 89.7
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Participants Achieving an sPGA (0) (Efficacy of Ixekizumab in Participants With Moderate to Severe Chronic Plaque Psoriasis. Measure: [sPGA])
Description: The sPGA is the physician's determination of the participant's Ps lesions overall at a given time point. Lesions were categorized by descriptions for induration, erythema, and scaling. Participant's Ps was assessed as 0 (clear), 1 (minimal), 2 (mild), 3 (moderate), 4 (severe), or 5 (very severe).
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 168 | 358 | 347 | 351
percentage of participants | 0.6 | 5.9 | 32.3 | 41.9
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

4. Secondary Outcome: Percentage of Participants Achieving PASI 90% (PASI90) (Efficacy of Ixekizumab in Participants With Moderate to Severe Chronic Plaque Psoriasis. Measure: [PASI])
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores were then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor (head [0.1], upper limbs [0.2], trunk [0.3], lower limbs [0.4]). Overall scores range from 0 (no Ps) to 72 (the most severe disease). Participants achieving PASI90 were defined as having an improvement of ≥90% in the PASI score compared to baseline.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 168 | 358 | 347 | 351
percentage of participants | 0.6 | 18.7 | 59.7 | 70.7
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

5. Secondary Outcome: Percentage of Participants Achieving PASI 100% (PASI100)
Description: The PASI combines the extent of body surface involvement in 4 anatomical regions (head, trunk, arms, and legs). For each region the percent area of skin involved was estimated from 0 (0%) to 6 (90%-100%) and severity was estimated by clinical signs of erythema, induration and scaling with a scores range from 0 (no involvement) to 4 (severe involvement). Each area is scored by itself and the scores were then combined for the final PASI. Final PASI calculated as: sum of severity parameters for each region * area score * weighing factor (head [0.1], upper limbs [0.2], trunk [0.3], lower limbs [0.4]). Overall scores range from 0 (no Ps) to 72 (the most severe disease). Participants achieving PASI100 were defined as having an improvement of 100% in the PASI score compared to baseline.
Time Frame: Week 12
Population: All randomized participants. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for NRI analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 168 | 358 | 347 | 351
percentage of participants | 0.6 | 5.3 | 30.8 | 40.5
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Test type: Superiority or Other; p = 0.008, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

6. Secondary Outcome: Percentage of Participants Maintaining an sPGA (0,1) From Week 12 After Re-randomization at Start of Maintenance Dosing Period to Week 60
Description: as for outcome 3
Time Frame: Week 60
Population: All randomized participants who had sPGA score of (0,1) at Week 12, were re-randomized at Week 12 and received at least 1 dose of study treatment in the Maintenance Dosing Period. Participants who did not meet the clinical response criteria or had missing data at Week 60 were considered non-responders for Non-Responder Imputation (NRI) analysis.
Measure: Number; unit: Percentage of participants
Groups:
- Ixe/Placebo- Maintenance Period Primary Pop: Participants who received 80 mg ixe Q2W or Q4W in Induction Period (Weeks 0 to 10) and classified as responders were administered placebo as 2 SC injections at Week 12 followed by placebo as 1 SC injection Q4W up to and including Week 56.
Arm/Group | Ixe/Placebo- Maintenance Period Primary Pop | Ixe/Ixe Q12W - Maintenance Period Primary Pop | Ixe/Ixe Q4W - Maintenance Period Primary Pop
Number analyzed (Participants) | 176 | 181 | 187
Percentage of participants | 6.3 | 40.9 | 74.9
Statistical Analysis 1: Comparison: Ixe/Placebo- Maintenance Period Primary Pop vs Ixe/Ixe Q12W - Maintenance Period Primary Pop; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Ixe/Placebo- Maintenance Period Primary Pop vs Ixe/Ixe Q4W - Maintenance Period Primary Pop; Test type: Superiority or Other; p < 0.001, Fisher Exact

7. Secondary Outcome: Percentage of Participants With Itching Severity (Itch Numeric Rating Scale [NRI]) Score ≥4 Point Reduction From Baseline
Description: The Itch Numeric Rating Scale (NRS) is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable". The number and percentage of participants achieving an Itch NRS ≥4 point reduction from baseline were presented by treatment group for participants who had a baseline Itch NRS ≥4. Describes worst level of itching in past 24 hours.
Time Frame: Week 12
Population: All randomized participants who had Itch NRS ≥4 at baseline. Participants who did not meet the clinical response criteria or had missing data at Week 12 were considered non-responders for NRI analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 135 | 306 | 293 | 303
percentage of participants | 14.1 | 57.8 | 76.8 | 85.1
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

8. Secondary Outcome: Change From Baseline in Dermatology-Specific Quality of Life Index (DLQI) Total Score (Quality of Life and Outcome Assessments. Measures: Participant Reported Outcomes [PRO])
Description: DLQI is a participant-administered, 10-question, validated, quality-of-life questionnaire that covers 6 domains, including symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include 0 (not at all), 1 (a little), 2 (a lot), and 3 (very much); and "not relevant" and unanswered responses were scored as "0." Total scores range from 0 to 30, with higher score indicating greater quality of life impairment. A 5-point change from baseline is considered clinically relevant. Least Squares (LS) Mean change from baseline was calculated using mixed model repeated measures (MMRM) with baseline score as covariate, treatment, pooled center, visit and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who had baseline and at least 1 post-baseline DLQI measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 160 | 346 | 338 | 343
units on a scale | -2.0 (0.36) | -7.7 (0.25) | -9.4 (0.25) | -10.4 (0.25)
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

9. Secondary Outcome: Change From Baseline in Nail Psoriasis Severity Index (NAPSI)
Description: The NAPSI scale is used to evaluate the severity of fingernail bed Ps and fingernail matrix Ps. The fingernail bed and fingernail matrix are each divided into quadrants. Each fingernail is given a score for fingernail bed Ps and fingernail matrix Ps, each with scores of 0 (none) to 4 (Ps in all 4 quadrants), depending on the presence (score of 1) or absence (score of 0) of Ps in each quadrant of the fingernail bed or matrix. The NAPSI score of a fingernail is the sum of scores from each quadrant of the fingernail bed and fingernail matrix (maximum of 8). The total NAPSI score equals the sum of all fingernails and ranges from 0 to 80 with higher scores indicating more severe Ps. LS mean change from baseline in NAPSI score was calculated using MMRM with baseline score as covariate, treatment, pooled center, visit and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who had fingernail Ps involvement at baseline and at least 1 post-baseline NAPSI measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 111 | 219 | 215 | 206
units on a scale | -0.82 (1.162) | -5.34 (0.835) | -7.39 (0.843) | -8.60 (0.853)
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

10. Secondary Outcome: Change From Baseline Psoriasis Scalp Severity Index (PSSI) Score
Description: The PSSI is a physician assessment of erythema, induration and desquamation and percent of scalp that is covered with a scores range from 0 (none) to 4 (very severe). The composite score is derived from the sum of scores for erythema, induration, and desquamation multiplied by the score recorded for the extent of the scalp area involved, 1 (<10%) to 6 (90%-100%) with a total scores range from 0 (less severity) to 72 (more severity), with lower scores indicating less severity. LS mean change from baseline in PSSI score was calculated using MMRM with baseline score as a covariate, treatment, pooled center, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who had scalp Ps involvement at baseline and at least 1 post-baseline PSSI measurement. Missing data was imputed by last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 150 | 316 | 307 | 318
units on a scale | -3.8 (0.73) | -14.8 (0.50) | -18.5 (0.51) | -18.7 (0.50)
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

11. Secondary Outcome: Change From Baseline in Percent of Body Surface Area (BSA) Involvement of Psoriasis
Description: The percentage involvement of psoriasis on each participant's body surface area was assessed by the investigator on a continuous scale from 0% (no involvement) to 100% (full involvement), in which 1% corresponds to the size of the participant's hand including palm, fingers and thumb. LS mean change from baseline in BSA was calculated using MMRM with baseline BSA as a covariate, treatment, pooled center, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, Week 12
Population: All randomized participants who had at least 1 post-baseline BSA measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 166 | 350 | 342 | 348
units on a scale | 0.5 (1.05) | -12.4 (0.72) | -20.3 (0.72) | -20.6 (0.71)
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

12. Secondary Outcome: Change From Baseline in Quick Inventory of Depressive Symptomatology-Self Report 16 Items (QIDS-SR16) Total Score
Description: The QIDS-SR16 is a self-administered, 16-item instrument in which a participant is asked to consider each statement as it relates to the way they have felt for the past 7 days. There is a 4-point scale for each item ranging from 0 (best) to 3 (worst). The 16 items are scored to give 9 individual depression domains (sad mood, concentration, self-criticism, suicidal ideation, interest, energy/fatigue, sleep disturbance [initial, middle and late insomnia or hypersomnia], decrease/increase in appetite/weight, and psychomotor agitation/retardation), which are summed to give a single score ranging from 0 to 27, with higher scores denoting greater symptom severity. LS mean change from baseline in total QIDS-SR16 score was calculated using the analysis of covariance (ANCOVA) model with treatment, pooled center and baseline QIDS total score.
Time Frame: Baseline, Week 12
Population: All randomized participants who had baseline and at least 1 post baseline QIDS-SR16 measurement. Missing data was imputed by last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 162 | 342 | 334 | 347
units on a scale | 0.1 (0.21) | -0.3 (0.15) | -0.7 (0.15) | -0.9 (0.15)
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Test type: Superiority or Other; p = 0.150, ANCOVA
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Test type: Superiority or Other; p = 0.002, ANCOVA
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Test type: Superiority or Other; p < 0.001, ANCOVA

13. Secondary Outcome: Change From Baseline in All Scores of the Work Productivity Activity Impairment Questionnaire-Psoriasis (WPAI-PSO)
Description: The (WPAI-PSO) is a 6-item instrument used to assess the impact of psoriasis on productivity impairment within the past 7 days and has four domains, namely, absenteeism, presenteeism (reduced productivity while at work), an overall work impairment score, and impairment in daily activities performed outside of work. Four scores are derived as percentages: absenteeism, presenteeism, overall work impairment (absenteeism and presenteeism), and impairment in activities performed outside of work. Percentage is calculated as each score * 100 and ranges from 0 to 100; greater scores indicate greater impairment. LS mean change from baseline in each WPAI-PSO score was calculated using the (ANCOVA) model with treatment, pooled center and baseline WPAI value.
Time Frame: Baseline, Week 12
Population: All randomized participants who had baseline and at least 1 post baseline WPAI-PSO measurement. Missing data was imputed by last observation carried forward ( LOCF ).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 160 | 342 | 332 | 340
units on a scale
  Absenteeism: number analyzed (Participants) | 87 | 199 | 204 | 213
  Absenteeism | -1.5 (0.83) | -3.7 (0.55) | -3.2 (0.54) | -3.9 (0.54)
  Activity Impairment Score | -0.4 (1.46) | -16.6 (1.00) | -22.6 (1.02) | -25.8 (1.01)
  Presenteeism Score: number analyzed (Participants) | 94 | 217 | 226 | 232
  Presenteeism Score | -2.4 (1.59) | -12.4 (1.05) | -18.5 (1.03) | -18.2 (1.03)
  Work Productivity Loss Score: number analyzed (Participants) | 86 | 199 | 203 | 211
  Work Productivity Loss Score | -2.0 (1.80) | -13.7 (1.18) | -19.3 (1.18) | -19.5 (1.18)
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Absenteeism Score; Test type: Superiority or Other; p = 0.026, ANCOVA
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Absenteeism Score; Test type: Superiority or Other; p = 0.076, ANCOVA
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Absenteeism Score; Test type: Superiority or Other; p = 0.016, ANCOVA
Statistical Analysis 4: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Activity Impairment Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 5: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Activity Impairment Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 6: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Activity Impairment Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 7: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Presenteeism Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 8: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Presenteeism Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 9: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Presenteeism Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 10: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Work Productivity Loss Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 11: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Work Productivity Loss Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 12: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Work Productivity Loss Score; Test type: Superiority or Other; p < 0.001, ANCOVA

14. Secondary Outcome: Change From Baseline in Medical Outcomes Study 36-Item Short Form Health Survey (SF-36) and Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores
Description: The SF-36 is a participant-reported outcome measure evaluating participant's health status. It comprises 36 items covering 8 domains: physical functioning, role physical, role emotional, bodily pain, vitality, social functioning, mental health, and general health. Items are answered on Likert scales of varying lengths. The 8 domains are regrouped into the PCS and MCS scores. The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health. In this study, the SF-36 acute version was used, which has a 1 week recall period. LS mean change from baseline in SF-36 score was calculated using the ANCOVA model with treatment, pooled center and baseline SF-36 score.
Time Frame: Baseline, Week 12
Population: All randomized participants who had baseline and at least 1 post baseline SF-36 measurement. Missing data was imputed by last observation carried forward ( LOCF ).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 158 | 336 | 333 | 344
units on a scale
  Physical Summary Score | -0.4495 (0.5226) | 2.5498 (0.3610) | 4.5726 (0.3628) | 3.7964 (0.3575)
  Mental Summary Score | -0.0955 (0.5886) | 2.3221 (0.4065) | 2.8504 (0.4090) | 4.5142 (0.4026)
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Physical Summary Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Physical Summary Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Physical Summary Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 4: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Mental Summary Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 5: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Mental Summary Score; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 6: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Mental Summary Score; Test type: Superiority or Other; p < 0.001, ANCOVA

15. Secondary Outcome: Change From Baseline in Patient's Global Assessment (PatGA) of Disease Severity
Description: The Patient's Global Assessment of Disease Severity is a single-item patient reported outcome measure on which participants are asked to rate by circling a number on a 0 to 5 NRS the severity of their psoriasis "today" from 0 (Clear) = no psoriasis to 5 (Severe) = the worst their psoriasis has ever been. LS mean change from baseline in patient's global assessment of disease severity score was calculated using (MMRM) with baseline score as a covariate, treatment, pooled center, visit, and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline, 12 weeks
Population: All randomized participants who had baseline and at least 1 post baseline PatGA measurement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 164 | 348 | 339 | 343
units on a scale | -0.4 (0.09) | -2.1 (0.06) | -3.0 (0.06) | -3.2 (0.06)
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

16. Secondary Outcome: Percentage of Participants Achieving Palmoplantar PASI (PPASI) of ≥50% (PPASI50), ≥75% (PPASI75) or 100% (PPASI100) Improvement
Description: The Palmoplantar PASI is a composite score derived from the sum scores for erythema, induration, and desquamation multiplied by a score for the extent of palm and sole area involvement, ranging from 0 to 72. The PPASI was only assessed if participants have palmoplantar psoriasis at baseline. Participants achieving PPASI50, PPASI75 or PASI100 were defined as having an improvement of at least 50%, 75%, or of 100%, respectively, in the PPASI scores compared to baseline.
Time Frame: Week 12
Population: All randomized participants who had palmoplantar Ps involvement at baseline. Participants who did not meet clinical response criteria or have missing data will be considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 55 | 95 | 102 | 104
percentage of participants
  PPASI 50 | 43.6 | 71.6 | 85.3 | 88.5
  PPASI 75 | 30.9 | 61.1 | 80.4 | 79.8
  PPASI 100 | 25.5 | 50.5 | 69.6 | 71.2
Statistical Analysis 1: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; PPASI 50; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; PPASI 50; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; PPASI 50; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; PPASI 75; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; PPASI 75; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 6: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; PPASI 75; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 7: Comparison: Placebo - Induction Period vs 50 mg ETN - Induction Period; PPASI 100; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel
Statistical Analysis 8: Comparison: Placebo - Induction Period vs Ixe Q4W - Induction Period; PPASI 100; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel
Statistical Analysis 9: Comparison: Placebo - Induction Period vs Ixe Q2W - Induction Period; PPASI 100; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel

17. Secondary Outcome: Percentage of Participants With Anti-Ixekizumab Antibodies
Description: Percentage of participants with treatment-emergent positive anti-ixekizumab antibodies was summarized by treatment group. Percentage was calculated based on the # of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-ixekizumab antibodies / number of evaluable participants * 100%.
Time Frame: Baseline to Week 12
Population: All randomized participants who received at least 1 dose of study treatment and had evaluable data.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period
Number analyzed (Participants) | 165 | 347 | 340 | 346
percentage of participants | 0 | 2.9 | 14.1 | 10.4

ADVERSE EVENTS:
Time Frame: Up to 288 Weeks
Description: Adverse events were summarized based on all randomized participants who received at least one dose of study treatment. The gender specific events only occurring in male or female participants were adjusted accordingly.
Groups:
- Ixe Q4W - Induction Period: 160 mg ixe was administered as 2 SC injections at Week 0 followed by 80 mg ixe as 1 SC injection every 4 weeks (Q4W): (Weeks 4 and 8). Placebo was administered as 1 SC injection at Weeks 2, 6, and 10. Placebo for ETN (1 SC injection) was administered twice weekly starting at Week 0 up to Week 12.
- Placebo Resp/Placebo - Maintenance Period Secondary Pop: Participants who received placebo during the Induction Period (Weeks 0 to 10) and classified as responders and were administered placebo as 2 SC injections at Week 12 followed by placebo as 1 SC injection Q4W up to and including Week 56.
- Placebo NonResp/Ixe Q4W - Maintenance Period Secondary Pop: Participants who received placebo in Induction Period (Weeks 0 to 10) and classified as non-responders were administered 160 mg ixe as 2 SC injections at Week 12 followed by 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- Ixe Q4W NonResp/Ixe Q4W- Maintenance Period Secondary Pop: Participants who received 80 mg ixe Q4W in Induction Period (Weeks 0 to 10) and classified as non-responders were administered 80 mg ixe as 1 SC injection and a Placebo for ixe injection at Week 12 followed by 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- Ixe Q2W NonResp/Ixe Q4W Maintenance Period Secondary Pop: Participants who received 80 mg ixe Q2W in Induction Period (Weeks 0 to 10) and classified as non-responders were administered 80 mg ixe as 1 SC injection and a Placebo for ixe injection at Week 12 followed by 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- Ixe Q4W Maintenance Period Relapsed Pop: Participants who relapsed (loss of response, sPGA ≥3 during Maintenance Period) were administered 80 mg ixe as 1 SC injection Q4W up to and including Week 56.
- Placebo Long-Term Extension: Participants who received placebo at the start of long-term extension period (Week 60) and could be switched to ixe. Data while participants were on placebo were included.
Arm/Group | Placebo - Induction Period | 50 mg ETN - Induction Period | Ixe Q4W - Induction Period | Ixe Q2W - Induction Period | Ixe/Placebo- Maintenance Period Primary Pop | Ixe/Ixe Q4W - Maintenance Period Primary Pop | Ixe/Ixe Q12W - Maintenance Period Primary Pop | Placebo Resp/Placebo - Maintenance Period Secondary Pop | Placebo NonResp/Ixe Q4W - Maintenance Period Secondary Pop | ETN Resp/Placebo Maintenance Period Secondary Pop | ETN NonResp/Ixe Q4W - Maintenance Period Secondary Pop | Ixe Q4W NonResp/Ixe Q4W- Maintenance Period Secondary Pop | Ixe Q2W NonResp/Ixe Q4W Maintenance Period Secondary Pop | Ixe Q4W Maintenance Period Relapsed Pop | Placebo Long-Term Extension | Ixe Long-Term Extension | Total Ixe Long-Term Extension | Placebo Post-Treatment Follow-Up | ETN Post-Treatment Follow-Up | Ixe Q2W Post-Treatment Follow-Up | Ixe Q4W Post-Treatment Follow-Up | Ixe Q12W Post-Treatment Follow-Up
Serious Adverse Events (participants affected / at risk) | 3/167 | 8/357 | 8/347 | 5/350 | 8/176 | 12/187 | 14/181 | 0/3 | 13/155 | 2/132 | 9/200 | 4/75 | 2/49 | 14/368 | 1/26 | 107/979 | 107/1002 | 1/16 | 0/6 | 3/248 | 12/656 | 0/24
Other Adverse Events (participants affected / at risk) | 48/167 | 141/357 | 116/347 | 140/350 | 56/176 | 100/187 | 87/181 | 2/3 | 77/155 | 42/132 | 106/200 | 27/75 | 26/49 | 136/368 | 7/26 | 345/979 | 345/1002 | 2/16 | 3/6 | 21/248 | 34/656 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Induction Period (N=167) | 50 mg ETN - Induction Period (N=357) | Ixe Q4W - Induction Period (N=347) | Ixe Q2W - Induction Period (N=350) | Ixe/Placebo- Maintenance Period Primary Pop (N=176) | Ixe/Ixe Q4W - Maintenance Period Primary Pop (N=187) | Ixe/Ixe Q12W - Maintenance Period Primary Pop (N=181) | Placebo Resp/Placebo - Maintenance Period Secondary Pop (N=3) | Placebo NonResp/Ixe Q4W - Maintenance Period Secondary Pop (N=155) | ETN Resp/Placebo Maintenance Period Secondary Pop (N=132) | ETN NonResp/Ixe Q4W - Maintenance Period Secondary Pop (N=200) | Ixe Q4W NonResp/Ixe Q4W- Maintenance Period Secondary Pop (N=75) | Ixe Q2W NonResp/Ixe Q4W Maintenance Period Secondary Pop (N=49) | Ixe Q4W Maintenance Period Relapsed Pop (N=368) | Placebo Long-Term Extension (N=26) | Ixe Long-Term Extension (N=979) | Total Ixe Long-Term Extension (N=1002) | Placebo Post-Treatment Follow-Up (N=16) | ETN Post-Treatment Follow-Up (N=6) | Ixe Q2W Post-Treatment Follow-Up (N=248) | Ixe Q4W Post-Treatment Follow-Up (N=656) | Ixe Q12W Post-Treatment Follow-Up (N=24)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frenulum breve (Congenital, familial and genetic disorders) | 0/119 (0) | 0/235 (0) | 0/244 (0) | 0/221 (0) | 0/110 (0) | 0/131 (0) | 0/120 (0) | 0/1 (0) | 0/112 (0) | 0/89 (0) | 0/126 (0) | 0/53 (0) | 0/30 (0) | 0/239 (0) | 0/14 (0) | 1/666 (1) | 1/678 (1) | 0/10 (0) | 0/5 (0) | 0/170 (0) | 0/453 (0) | 0/14 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic ischaemic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrophic anal papilla (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Noninfective sialoadenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal achalasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyp (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bartholin's abscess (Infections and infestations) | 0/48 (0) | 0/122 (0) | 0/103 (0) | 0/129 (0) | 0/66 (0) | 0/56 (0) | 0/61 (0) | 0/2 (0) | 0/43 (0) | 0/43 (0) | 0/74 (0) | 0/22 (0) | 0/19 (0) | 1/129 (1) | 0/12 (0) | 0/313 (0) | 0/324 (0) | 0/6 (0) | 0/1 (0) | 0/78 (0) | 0/203 (0) | 0/10 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (8) | 6 (8) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema infected (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 0/48 (0) | 0/122 (0) | 0/103 (0) | 0/129 (0) | 0/66 (0) | 0/56 (0) | 0/61 (0) | 0/2 (0) | 0/43 (0) | 0/43 (0) | 0/74 (0) | 0/22 (0) | 0/19 (0) | 0/129 (0) | 0/12 (0) | 1/313 (1) | 1/324 (1) | 0/6 (0) | 0/1 (0) | 0/78 (0) | 0/203 (0) | 0/10 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exposure via father (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0/48 (0) | 0/122 (0) | 0/103 (0) | 0/129 (0) | 0/66 (0) | 0/56 (0) | 0/61 (0) | 0/2 (0) | 0/43 (0) | 0/43 (0) | 0/74 (0) | 0/22 (0) | 0/19 (0) | 0/129 (0) | 0/12 (0) | 1/313 (1) | 1/324 (1) | 0/6 (0) | 0/1 (0) | 0/78 (0) | 0/203 (0) | 0/10 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mycobacterium tuberculosis complex test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/119 (0) | 0/235 (0) | 0/244 (0) | 0/221 (0) | 0/110 (0) | 1/131 (1) | 1/120 (1) | 0/1 (0) | 0/112 (0) | 0/89 (0) | 0/126 (0) | 0/53 (0) | 0/30 (0) | 0/239 (0) | 0/14 (0) | 3/666 (3) | 3/678 (3) | 0/10 (0) | 0/5 (0) | 0/170 (0) | 0/453 (0) | 0/14 (0)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/48 (0) | 0/122 (0) | 0/103 (0) | 0/129 (0) | 1/66 (1) | 0/56 (0) | 0/61 (0) | 0/2 (0) | 0/43 (0) | 0/43 (0) | 0/74 (0) | 0/22 (0) | 0/19 (0) | 0/129 (0) | 0/12 (0) | 0/313 (0) | 0/324 (0) | 0/6 (0) | 0/1 (0) | 0/78 (0) | 0/203 (0) | 0/10 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/48 (0) | 0/122 (0) | 0/103 (0) | 0/129 (0) | 0/66 (0) | 0/56 (0) | 0/61 (0) | 0/2 (0) | 0/43 (0) | 0/43 (0) | 0/74 (0) | 0/22 (0) | 0/19 (0) | 1/129 (1) | 0/12 (0) | 1/313 (1) | 1/324 (1) | 0/6 (0) | 0/1 (0) | 0/78 (0) | 1/203 (1) | 0/10 (0)
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 0/48 (0) | 0/122 (0) | 0/103 (0) | 0/129 (0) | 0/66 (0) | 0/56 (0) | 0/61 (0) | 0/2 (0) | 1/43 (1) | 0/43 (0) | 0/74 (0) | 0/22 (0) | 0/19 (0) | 0/129 (0) | 0/12 (0) | 0/313 (0) | 0/324 (0) | 0/6 (0) | 0/1 (0) | 0/78 (0) | 0/203 (0) | 0/10 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Schizophrenia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acquired hydrocele (Reproductive system and breast disorders) | 0/119 (0) | 0/235 (0) | 0/244 (0) | 0/221 (0) | 0/110 (0) | 0/131 (0) | 0/120 (0) | 0/1 (0) | 0/112 (0) | 0/89 (0) | 0/126 (0) | 0/53 (0) | 0/30 (0) | 0/239 (0) | 0/14 (0) | 1/666 (1) | 1/678 (1) | 0/10 (0) | 0/5 (0) | 0/170 (0) | 0/453 (0) | 0/14 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/119 (0) | 0/235 (0) | 0/244 (0) | 0/221 (0) | 0/110 (0) | 0/131 (0) | 0/120 (0) | 0/1 (0) | 0/112 (0) | 0/89 (0) | 0/126 (0) | 0/53 (0) | 0/30 (0) | 0/239 (0) | 0/14 (0) | 2/666 (2) | 2/678 (2) | 0/10 (0) | 0/5 (0) | 0/170 (0) | 0/453 (0) | 0/14 (0)
Penile dysplasia (Reproductive system and breast disorders) | 0/119 (0) | 0/235 (0) | 0/244 (0) | 0/221 (0) | 0/110 (0) | 0/131 (0) | 0/120 (0) | 0/1 (0) | 0/112 (0) | 0/89 (0) | 0/126 (0) | 0/53 (0) | 0/30 (0) | 0/239 (0) | 0/14 (0) | 1/666 (3) | 1/678 (3) | 0/10 (0) | 0/5 (0) | 0/170 (0) | 0/453 (0) | 0/14 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine dilation and curettage (Surgical and medical procedures) | 0/48 (0) | 0/122 (0) | 0/103 (0) | 0/129 (0) | 0/66 (0) | 0/56 (0) | 0/61 (0) | 0/2 (0) | 0/43 (0) | 0/43 (0) | 0/74 (0) | 0/22 (0) | 0/19 (0) | 0/129 (0) | 0/12 (0) | 0/313 (0) | 0/324 (0) | 0/6 (0) | 0/1 (0) | 1/78 (1) | 0/203 (0) | 0/10 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic dilatation (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo - Induction Period (N=167) | 50 mg ETN - Induction Period (N=357) | Ixe Q4W - Induction Period (N=347) | Ixe Q2W - Induction Period (N=350) | Ixe/Placebo- Maintenance Period Primary Pop (N=176) | Ixe/Ixe Q4W - Maintenance Period Primary Pop (N=187) | Ixe/Ixe Q12W - Maintenance Period Primary Pop (N=181) | Placebo Resp/Placebo - Maintenance Period Secondary Pop (N=3) | Placebo NonResp/Ixe Q4W - Maintenance Period Secondary Pop (N=155) | ETN Resp/Placebo Maintenance Period Secondary Pop (N=132) | ETN NonResp/Ixe Q4W - Maintenance Period Secondary Pop (N=200) | Ixe Q4W NonResp/Ixe Q4W- Maintenance Period Secondary Pop (N=75) | Ixe Q2W NonResp/Ixe Q4W Maintenance Period Secondary Pop (N=49) | Ixe Q4W Maintenance Period Relapsed Pop (N=368) | Placebo Long-Term Extension (N=26) | Ixe Long-Term Extension (N=979) | Total Ixe Long-Term Extension (N=1002) | Placebo Post-Treatment Follow-Up (N=16) | ETN Post-Treatment Follow-Up (N=6) | Ixe Q2W Post-Treatment Follow-Up (N=248) | Ixe Q4W Post-Treatment Follow-Up (N=656) | Ixe Q12W Post-Treatment Follow-Up (N=24)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 6 (7) | 4 (5) | 4 (4) | 6 (8) | 0 (0) | 6 (6) | 1 (1) | 5 (5) | 1 (1) | 3 (4) | 5 (5) | 1 (1) | 20 (21) | 20 (21) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (6) | 1 (2) | 5 (6) | 7 (7) | 2 (3) | 2 (2) | 4 (4) | 0 (0) | 6 (7) | 2 (2) | 4 (6) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 11 (11) | 11 (11) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 2 (2) | 18 (64) | 9 (10) | 12 (20) | 2 (3) | 3 (6) | 4 (4) | 0 (0) | 5 (14) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 5 (19) | 5 (19) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (33) | 4 (5) | 5 (33) | 13 (79) | 4 (22) | 1 (3) | 1 (13) | 0 (0) | 1 (5) | 1 (1) | 2 (4) | 0 (0) | 1 (2) | 1 (1) | 1 (18) | 1 (21) | 1 (21) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 38 (192) | 19 (30) | 40 (76) | 0 (0) | 15 (69) | 4 (8) | 0 (0) | 10 (42) | 1 (3) | 20 (80) | 3 (21) | 2 (2) | 19 (62) | 0 (0) | 21 (404) | 21 (404) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 5 (5) | 4 (4) | 5 (5) | 3 (3) | 7 (8) | 10 (12) | 0 (0) | 2 (2) | 0 (0) | 10 (11) | 1 (1) | 2 (3) | 11 (11) | 1 (1) | 38 (52) | 38 (52) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 12 (15) | 12 (15) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 17 (21) | 37 (41) | 28 (40) | 34 (34) | 19 (22) | 32 (42) | 24 (31) | 0 (0) | 29 (42) | 19 (24) | 35 (47) | 12 (13) | 8 (11) | 41 (61) | 0 (0) | 125 (195) | 125 (195) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 5 (5) | 5 (5) | 4 (4) | 1 (1) | 11 (12) | 3 (3) | 0 (0) | 3 (7) | 1 (1) | 7 (7) | 2 (2) | 4 (5) | 11 (13) | 0 (0) | 19 (26) | 19 (26) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 4 (4) | 6 (6) | 2 (2) | 3 (3) | 10 (10) | 6 (6) | 0 (0) | 7 (7) | 1 (1) | 7 (7) | 1 (1) | 0 (0) | 12 (12) | 0 (0) | 38 (56) | 38 (56) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (8) | 27 (27) | 16 (19) | 20 (21) | 14 (19) | 25 (30) | 21 (23) | 0 (0) | 20 (23) | 8 (9) | 21 (28) | 7 (10) | 7 (9) | 21 (32) | 2 (4) | 108 (166) | 108 (166) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 7 (7) | 5 (5) | 3 (3) | 5 (9) | 7 (9) | 1 (1) | 8 (8) | 0 (0) | 8 (14) | 1 (1) | 3 (3) | 4 (5) | 1 (1) | 27 (30) | 27 (30) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/48 (0) | 1/122 (1) | 0/103 (0) | 0/129 (0) | 1/66 (1) | 0/56 (0) | 0/61 (0) | 0/2 (0) | 1/43 (1) | 0/43 (0) | 2/74 (2) | 2/22 (2) | 0/19 (0) | 1/129 (1) | 0/12 (0) | 3/313 (3) | 3/324 (3) | 0/6 (0) | 0/1 (0) | 0/78 (0) | 0/203 (0) | 0/10 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 16 (17) | 16 (17) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mycobacterium tuberculosis complex test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 9 (10) | 8 (10) | 6 (6) | 5 (6) | 8 (10) | 10 (11) | 0 (0) | 6 (7) | 8 (10) | 10 (11) | 1 (1) | 1 (1) | 13 (14) | 0 (0) | 48 (60) | 48 (60) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (7) | 2 (2) | 4 (4) | 1 (2) | 9 (10) | 6 (8) | 0 (0) | 9 (9) | 2 (7) | 6 (6) | 3 (3) | 3 (3) | 12 (15) | 1 (1) | 40 (50) | 40 (50) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 5 (6) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 21 (22) | 17 (21) | 17 (23) | 7 (9) | 12 (14) | 8 (10) | 0 (0) | 8 (14) | 5 (6) | 4 (17) | 4 (4) | 4 (7) | 12 (19) | 0 (0) | 30 (46) | 30 (46) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 0/48 (0) | 0/122 (0) | 0/103 (0) | 0/129 (0) | 0/66 (0) | 1/56 (1) | 0/61 (0) | 0/2 (0) | 0/43 (0) | 0/43 (0) | 0/74 (0) | 0/22 (0) | 0/19 (0) | 0/129 (0) | 1/12 (1) | 2/313 (2) | 2/324 (2) | 0/6 (0) | 0/1 (0) | 0/78 (0) | 0/203 (0) | 0/10 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (7) | 5 (5) | 5 (5) | 1 (2) | 3 (3) | 5 (5) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 3 (4) | 7 (7) | 0 (0) | 12 (15) | 12 (15) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7) | 6 (6) | 5 (5) | 4 (4) | 3 (4) | 5 (6) | 0 (0) | 6 (8) | 2 (3) | 8 (10) | 3 (5) | 3 (3) | 12 (18) | 1 (1) | 28 (31) | 28 (31) | 0 (0) | 0 (0) | 3 (3) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days